CLINICAL TRIAL: NCT06487832
Title: Impact of the Incretin System on Brain Insulin Sensitivity in Humans with Normal Weight, Overweight and Obesity
Brief Title: Effect of GLP1 Receptor Agonist on Brain Insulin Responsiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 065/2024BO1
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Normal Weight; Overweight and Obesity; Insulin Sensitivity; Insulin Resistance
Keywords: GLP-1; Brain; functional magnetic resonance imaging; Semaglutide
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: In a randomized, single-blinded, within subject cross-over design, we will compare cerebral response from before to after intranasal insulin or placebo administration after a single dose of 0.25 mg semaglutide administration versus placebo administration
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 (Experimental): Acute administration of 0.25 mg semaglutide (0.19 ml)
  Interventions: Other: Subcutaneous GLP1-RA
- Placebo (Placebo Comparator): Acute administration of 0.19 ml NaCl
  Interventions: Other: Subcutaneous placebo

INTERVENTIONS:
Other: Subcutaneous GLP1-RA — Subcutaneous administration of semaglutide
  Arms: GLP-1
Other: Subcutaneous placebo — Subcutaneous administration of NaCl
  Arms: Placebo

SUMMARY:
The overarching goal of the current study is to investigate the effect of GLP-1 on brain insulin responsiveness in a randomized, single-blinded, within subject cross-over study design. To this end, investigators will compare the effect of the administration of semaglutide versus placebo, followed by an fMRI with administration of intranasal insulin or placebo.

DETAILED DESCRIPTION:
Investigate the effect of the GLP1 receptor agonist (i.e. 0.25 mg semaglutide) vs. placebo on the brain using functional magnetic resonance imaging (fMRI) in combination with 160IU intranasal insulin vs. placebo administration in healthy male and female participants of normal-weight and overweight/obesity. Participants will furthermore undergo tasks that assess cognitive functions and eating behavior. Brain insulin responsiveness (primary outcome) is defined as the cerebral response to intranasal insulin compared to placebo by means of cerebral blood flow and resting-state BOLD measurements. Secondary outcomes include diffusion weighted imaging, neural food cue reactivity, cognitive functions and metabolic predictors.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 24.9 kg/m2; and between 27.5 kg/m2 and 40 kg/m2
* Written consent to participate in the study
* Written consent to be informed about incidental findings

Exclusion Criteria:

* Type 1 or type 2 diabetes, LADA, MODY, or cardiovascular diseases such as chronic heart failure, myocardial infarction, status post stroke
* BMI < 18.5 or > 40 kg/m2
* Persons who cannot legally give consent
* Pregnancy or lactation
* History of severe mental or somatic disorders including neurological diseases (incl. epileptic seizures)
* Taking psychotropic drugs
* Chronic diseases or medication that influence glucose metabolism
* Regular use of analgesic drugs
* Previous bariatric surgery
* Known allergy against one or more of the used agents
* Acute infection and/or antibiotic treatment within the last 4 weeks
* Hemoglobin values less than 10.5 g/dl for women, less than 11.5 g/dl for men
* Other diseases that in the opinion of the investigator may jeopardize the success of the study or indicate a risk to the volunteer
* Participation in a lifestyle intervention study or a pharmaceutical study within the last 30 days
* Metal implants which cannot be removed as pacemakers, artificial heart valve, electrical devices as insulin pumps, large tattoos, retainer over more than 4 teeth, contraceptive coil, implanted magnetic metal parts as screws or plates after a surgery
* Persons with claustrophobia
* Persons with tinnitus
* Weight loss or gain of >5% in the last 3 months
* Pancreatic diseases
* History or family history of multiple endocrine neoplasia (MEN2) or medullary thyroid cancer
* History of malignant thyroid disease
* History of malignant disease in the past 5 years
* Surgery in the last three months
* Chronic tobacco use of more than 10 cigarettes/day
* Women who do not consent to refrain from breastfeeding until 2 months after the end of the study
* Women of childbearing age who do not consent to use safe method of contraception from 28 days before until 2 months after the end of the study or refrain from heterosexual intercourse during this time
* Women of childbearing age who do not consent to take a pregnancy test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral response after insulin compared to placebo nasal spray | 24 hours after semaglutide or placebo administration
  Resting-state cerebral blood flow and BOLD-fMRI response from before to 30 min after nasal spray administration

SECONDARY OUTCOMES:
Neural food-cue reactivity after insulin compared to placebo nasal spray | 24 hours after semaglutide or placebo administration
  BOLD-fMRI response to food cues 30 min after nasal spray administration
Diffusion-weighted imaging (DWI) | 24 hours after semaglutide or placebo administration
  Diffusion weighted parameter based on MRI measurements
Heart rate variability (HRV) | 24 hours after semaglutide or placebo administration
  HRV based on ECG measurements
Change in subjective feeling of hunger and food craving | 24 hours after semaglutide or placebo administration
  On a visual analogue scale, subjective feeling of hunger and food craving will be assessed using questionnaires.
Change in mood | 24 hours after semaglutide or placebo administration
  Using a questionnaire, positive and negative affect state will be assessed.
Performance during cognitive tests | 24 hours after semaglutide or placebo administration
  Cambridge Cognition Tests Battery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas L. Birkenfeld, MD, Study Director — Institute for Diabetes research and Metabolic Diseases at the University of Tubingen
Locations (1):
- University Clinic Tubingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No